CLINICAL TRIAL: NCT00352794
Title: Evaluation of Lenalidomide (CC-5013) and Prednisone as a Therapy for Patients With Myelofibrosis (MF)
Brief Title: Lenalidomide for Patients With Myelofibrosis (MF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0206
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Myelofibrosis
Keywords: Combination chemotherapy; Myelofibrosis (MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Lenalidomide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Prednisone (Experimental): Lenalidomide oral 10 mg daily/days 1-21 of 28 day cycle. Prednisone starting dose oral 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  Interventions: Drug: Lenalidomide; Drug: Prednisone

INTERVENTIONS:
Drug: Lenalidomide — Oral 10 mg daily/days 1-21 of 28 day cycle
Drug: Prednisone — Starting dose oral 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide in combination with prednisone can help to control myelofibrosis. The safety of lenalidomide and prednisone for the treatment of myelofibrosis will also be studied.

DETAILED DESCRIPTION:
Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells. Prednisone is designed to improve the results of lenalidomide and to help reduce the side effects.

If you are found to be eligible to take part in this study, you will take 1-2 capsules of lenalidomide by mouth daily. You will take lenalidomide daily for 21 days followed by 1 week rest. This 28-day period is called a study "cycle."

Swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

You will take prednisone by mouth every day during Cycles 1-2, and every other day during Cycle 3. You may only take prednisone for Cycles 1-3.

You will be given a study drug diary. In this diary, you will record when you take the study drug(s).

During treatment, blood (about 1 tablespoon) will be drawn once every 1-2 weeks. Following the completion of 24 cycles, blood (about 1 tablespoon) will be drawn every 1- 3 months. The tests may be repeated more frequently to check for side effects.

Every month for the first 3 months, and then every 3 months, until you complete 24 cycles, you will have a study visit. You will have a bone marrow biopsy/aspirate every 3 months. Lenalidomide will be provided to you as a monthly (28-day) supply.

Following the completion of Cycle 24, you will have a study visit every 6 months. You will have a bone marrow biopsy/aspirate every 12 months. Lenalidomide will be provided to you as a monthly (28-day) supply.

Depending on side effects and the activity of the study drug against the disease, your dose of the study drug may be increased or decreased.

You may stay on study for as long as you are benefitting. You will be taken off study if you are not or are no longer benefitting or intolerable side effects occur.

This is an investigational study. Lenalidomide and prednisone are both FDA approved and commercially available. Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of patients with transfusion-dependent anemia due to Low- or Intermediate-1-risk myelodysplastic syndromes associated with the chromosome 5 abnormality with or without other chromosome abnormalities. Lenalidomide is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy. Myelodysplastic syndrome (MDS) and Multiple Myeloma (MM) are cancers of the blood. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental. Prednisone is on the market for many different things but not specifically for Myelofibrosis. The use of these drugs in combination is considered investigational in this study. Up to 41 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of myelofibrosis requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate or high risk according to Lille scoring system (risk factors are: Hb < 10 g/dl, White blood count (WBC) < 4 or > 30 x 109/L; risk group: 0 factor(s) = low, 1 factor(s) = intermediate, 2 factor(s) = high) or with symptomatic splenomegaly
2. Understanding and voluntary signing an Institutional Review Board (IRB)-approved informed consent form.
3. Age >/= 18 years at the time of signing the informed consent.
4. Disease-free of prior malignancies for >/= 2-years with exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
6. Patients must have adequate organ function as demonstrated by the following: Total bilirubin </= 2.0 mg/dL (unless higher due to MF); Serum creatinine </= 2.0 mg/dL (unless higher due to MF); Absolute neutrophil count >/= 1 x 10^9/L; Alanine transaminase (ALT) </= 3 x upper limit of normal (unless higher due to MF).
7. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
8. Continuation of 7. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix J: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods
9. footnote to no 7. † A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
10. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

1. Use of any other standard (e.g. hydroxyurea, anagrelide, growth factors) or experimental drug or therapy within 28 days of starting lenalidomide and/or lack of recovery from all toxicity from previous therapy to grade 1 or better.
2. Known prior clinically relevant hypersensitivity reaction to thalidomide, including the development of erythema nodosum if characterized by a desquamating rash.
3. Prior therapy with lenalidomide.
4. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
5. Suspected Pregnancy. Pregnant or lactating females.
6. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
7. Known positive for HIV or infectious hepatitis, type A, B or C.
8. Known prior clinically relevant hypersensitivity to prednisone.
9. Participants with a heart rate (HR) of less than or equal to 50, as a HR less than 50 indicates underlying cardiac abnormalities.
10. Participants with prior history of thromboembolic disease (i.e.-deep venous thrombosis (DVT) or pulmonary embolism (PE)) within the last six months, as Lenalidomide has demonstrated a significantly increased risk of DVT or PE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07-07 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Quintas-Cardama A, Kantarjian HM, Manshouri T, Thomas D, Cortes J, Ravandi F, Garcia-Manero G, Ferrajoli A, Bueso-Ramos C, Verstovsek S. Lenalidomide plus prednisone results in durable clinical, histopathologic, and molecular responses in patients with myelofibrosis. J Clin Oncol. 2009 Oct 1;27(28):4760-6. doi: 10.1200/JCO.2009.22.6548. Epub 2009 Aug 31. PMID 19720904
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2006 - April 2007
Period: Overall Study
Arm/Group | Lenalidomide + Prednisone
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide + Prednisone
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Response (Complete and Partial Response + Hematological Improvement)
Description: Time to response defined as the time from start of therapy until the response criteria are fulfilled. Response duration defined as the time from response until relapse (progressive disease) or death.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide + Prednisone
Number analyzed (Participants) | 40
Participants | 14

ADVERSE EVENTS:
Time Frame: For at least 6 cycles, and up to 11 years
Arm/Group | Lenalidomide + Prednisone
All-Cause Mortality (participants affected / at risk) | 3/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Prednisone (N=40)
Abdominal Pain (General disorders) | 1 (1)
Back Pain (General disorders) | 1 (3)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Increased Transaminase (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Mitral Heart Valve Repair (Surgical and medical procedures) | 1 (1)
Stent Replacement (Surgical and medical procedures) | 1 (1)
West Nile Virus (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Prednisone (N=40)
Neutropenia (Blood and lymphatic system disorders) | 21 (33)
Anemia (Blood and lymphatic system disorders) | 15 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (11)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3)
fatigue (General disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 12 (14)
Infection (Infections and infestations) | 17 (24)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 4 (4)
Edema (Blood and lymphatic system disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Depression (Nervous system disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Increased Transaminase (Hepatobiliary disorders) | 2 (3)
Sweating (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Headache (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 4 (4)
Pain (General disorders) | 21 (27)
Decreased White Blood Count (Blood and lymphatic system disorders) | 22 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT00352794/Prot_SAP_000.pdf